CLINICAL TRIAL: NCT04910802
Title: Concomitant HPV Vaccination and HPV Screening for Rapid Elimination of HPV Infection and Cervical Cancer in Sweden
Brief Title: Concomitant HPV Vaccination and HPV Screening HPV Infection and Cervical Cancer in Sweden
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Miriam Elfström (Other Government)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Miriam Elfström, Chief development officer, Region Stockholm
Organization: Region Stockholm (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Catch-up vaccination
Record Dates: First submitted 2021-05-01; First posted 2021-06-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: HPV Infection; CIN 2/3; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: All women in the targeted age-range will be offered vaccination in conjunction with screening.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HPV-vaccination (Experimental): Women ages 22-26 will be offered concomitant vaccination (1 dose of Gardasil9) and HPV screening. A second dose of Gardasil9 will be administered 3 years later.
  Interventions: Biological: Gardasil9

INTERVENTIONS:
Biological: Gardasil9 — Concomitant vaccination and HPV screening. Gardasil9 will be administered using standard dosage. 1 dose at recruitment and the 2nd dose 3 years later.

SUMMARY:
The study aims to evaluate whether organised, concomitant HPV vaccination and HPV screening offered to all resident women aged 22-27 will result in a more rapid elimination of HPV infection in Sweden. This objective will be examined at the population level.

DETAILED DESCRIPTION:
In Sweden, 150 women die of and 550 women are diagnosed with cervical cancer each year. The average age at diagnosis is about 55 years and every third woman is under 40 years of age. World-wide, there half a million new cases of cervical cancer each year. The underlying cause of cervical cancer is a human papillomavirus (HPV), an infection that can be prevented by vaccination. The first-generation vaccine protects against HPV infection of the two types (16 and 18) that cause to about 70% of all cervical cancer. Since 2015, a second-generation vaccine (Gardasil 9, Sanofi Pasteur MSD SNC) has been available that provides protection against 9 HPV types of which 7 types (16, 18, 31, 33, 35, 45, 52 and 58) cause 90% of all cervical cancer.

In 2016, the World Health Organization (WHO) called on the countries of the world to eliminate cervical cancer as a public health problem. On 17 November 2020, all 194 WHO member states adopted a global strategy to increase the rate of elimination of cervical cancer. The strategy involves three main actions: vaccination, screening, and treatment. In Sweden, girls have been offered school-based vaccination against HPV with Gardasil 4 since 2012. Starting in the autumn of 2020, schoolboys have also been offered vaccination. Since 2019, the second-generation vaccine has been used in the school-based vaccination program. Sweden's vaccination strategy means that the virus will be eliminated among individuals born in 2007 and beyond. It will thus take another 20 years before Sweden can stop the infection in Sweden. Today, the infection continues to spread only among young adults. Studies have shown that vaccination up to age 26 can be effective and within the European Union, 10 out of 29 countries have a so-called catch-up on vaccination program targeting women over the age of 20 but such a catch-up has not been formally introduced in Sweden.

The overall goal is to investigate whether offering women ages 22-26 years vaccination with Gardasil 9 in connection with screening may involve a faster eradication of cervical cancer as a public health problem in Sweden. A regional pilot study will be conducted in 2021 followed by a subsequent scale-up to other regions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will include resident women within the age range of 22-26, who have not opted out of the screening program and who consent to participate in the study.

Women who respond to the invitation and attend screening will be screened with HPV testing by the current routine practise. Women who consent to participate will also be offered HPV vaccination. The HPV vaccine (Gardasil 9) will be offered regardless of whether the woman reports having had prior vaccination with a first-generation vaccine (Gardasil 4) and regardless of screening test result.

Exclusion Criteria:

1. Known history of severe allergic reaction or hypersensitivity to any of the components of the HPV vaccine.For GARDASIL 9: Amorphous aluminium hydroxyphosphate sulphate adjuvant, Sodium chloride, L-histidine, Polysorbate 80 or Sodium borate
2. Known history of immune-related disorders
3. Current acute severe febrile illness, except for minor infections such as a cold, mild upper respiratory infection or low-grade fever.
4. Administration of immunoglobulin or blood-derived products within 6 months prior to scheduled HPV vaccine first dose
5. Current pregnancy (reported)
6. Women with a total hysterectomy

Ages: 22 Years to 27 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender eligibility is based on the sex coded in the personal identification number used in civil society in Sweden
Enrollment: 150000 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV | Measured at recruitment.
  Overall and type-specific prevalence of HPV will be obtained from the routine HPV screening programs in the regions that offer HPV screening to this age group.
Prevalence of HPV | Measured 3 years after recruitment, at the second cervical screening attendance.
  Overall and type-specific prevalence of HPV will be obtained from the routine HPV screening programs in the regions that offer HPV screening to this age group.
Prevalence of HPV | Measure 6 years after recruitment, at the third cervical screening attendance.
  Overall and type-specific prevalence of HPV will be obtained from the routine HPV screening programs in the regions that offer HPV screening to this age group.

SECONDARY OUTCOMES:
Number of women with histopathologically confirmed cervical intraepithelial neoplasia grade 2, 3, or cervical cancer (CIN2+) | Measured at recruitment, and subsequently at 3 year intervals.
  CIN2+ measured through registry linkages, by HPV type in the lesion.
Consumption of resources | Measured at recruitment, and subsequently at 3 year intervals.
  Number of screening and treatment visits.
Number of women with obstetrical complications | Measured at recruitment, and subsequently at 3 year intervals.
  Obstetrical complications such as preterm births measured through registry linkages.
Number of women with cervical specimens found to be benign | Measured at recruitment, and subsequently at 3 year intervals.
  Treatments for cervical abnormalities, measured as excised cervical specimens, found to be benign. Measured through registry linkages.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD, PhD, Study Director — Karolinska University Hospital Laboratory
Locations (1):
- Cancer prevention, screening, and counseling unit, Regional Cancer Center of Stockholm-Gotland, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Documents related to the study can be shared. Data, once collected, will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: The study protocol and informed consent form are available. The SAP will be made available and the analytic code will be available once the first round of results have been analyzed.
Access Criteria: Data can be shared with other researchers upon written request. Possibilities to share the data on a digital platform will be investigated.

REFERENCES:
- [Derived] Arroyo Muhr LS, Gini A, Yilmaz E, Hassan SS, Lagheden C, Hultin E, Garcia Serrano A, Ure AE, Andersson H, Merino R, Elfstrom KM, Baussano I, Dillner J. Concomitant human papillomavirus (HPV) vaccination and screening for elimination of HPV and cervical cancer. Nat Commun. 2024 May 1;15(1):3679. doi: 10.1038/s41467-024-47909-x. PMID 38693149